CLINICAL TRIAL: NCT06969716
Title: Frequency of Fibromyalgia Syndrome in Elderly Patients Aged 80 and Above and Its Relationship With Detailed Geriatric Assessment Parameters
Brief Title: Frequency of Fibromyalgia Syndrome in Elderly Patients Aged 80 and Above and Its Relationship With Geriatric Parameters
Status: Recruiting | Type: Observational
Sponsor: Sultan 1. Murat State Hospital (Other Government)
Responsible Party: Principal Investigator, Alper Mengi, Associate Professor, Sultan 1. Murat State Hospital
Other Study IDs: 27/3/2025-Number:03/29
Record Dates: First submitted 2025-05-03; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Fibromyalgia; Old Age; Debility
MeSH Terms: conditions — Fibromyalgia; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly Patients: Age 80 and above
  Interventions: Other: Detailed geriatric assessment

INTERVENTIONS:
Other: Detailed geriatric assessment — The demographic characteristics of the patients, comorbid diseases, history and number of falls in the last 6 months will be questioned, and the thyroid stimulating hormone, calciferol, cobalamin, glycosylated hemoglobin, folic acid and glomerular filtration rate levels routinely requested from each patient in the last 3 months will be recorded. During the outpatient clinic application, the patients will undergo neurocognitive assessment, mood assessment, daily living activities assessment, balance and walking assessment, nutritional assessment and frailty assessment. The patients' handgrip strength from their dominant hand will be assessed with a hand dynamometer. The walking speed of the patients will be measured as the number of seconds it takes to walk 4 meters and recorded in seconds. All patients will be questioned about the presence of body pain with the numerical pain scale score and all patients will be evaluated for the presence of fibromyalgia syndrome.

SUMMARY:
The aim of this study was to determine the prevalence of fibromyalgia syndrome in patients aged 80 years and over and to examine the relationship between detailed geriatric assessment parameters and fibromyalgia syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age 80 and above
* Patients with complete detailed geriatric assessment parameters

Exclusion Criteria:

* Presence of neurodegenerative disease (dementia, parkinsonism)
* Immobilized patient
* Those who have had an acute illness (infection, fracture, cerebrovascular disease) in the last month
* Having psychotic disorders
* Having severe hearing loss

Min Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients aged 80 and over who are followed up from the healthy aging outpatient clinic of Edirne Sultan 1. Murat State Hospital geriatric clinic will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Presence of fibromyalgia syndrome | Baseline
  The presence of fibromyalgia will be evaluated using the 2016 American College of Rheumatology diagnostic criteria.

SECONDARY OUTCOMES:
Neurocognitive assessment | Baseline
  Neurocognitive assessment will be done with Mini Mental State Examination (MMSE). MMSE test is a short screening test with 11 questions and 30 points. MMSE is completed in approximately 10 minutes and evaluates orientation, memory, attention, calculation, recall, language, motor function and perception, visual-spatial abilities. 24-30 points is normal, 18-23 points is mild dementia, 17 and below is compatible with severe dementia.
Mood assessment | Baseline
  Mood assessment will be assessed with the Geriatric Depression Scale-short form (GDS-SF). GDS-SF consists of 15 questions that patients answer yes or no. Scoring is done as the number of yes answers, and the total depression score is calculated from the sum of the scores. Scores between 0-9 are considered "normal", scores between 10-19 are considered "mild depression", and scores between 20-30 are considered "severe depression".
Daily living activities | Baseline
  The assessment of daily living activities will be assessed with the Lawton-Brody Instrumental Activities of Daily Living Scale (IADLS). IADLS consists of 8 questions that include information on using the telephone, preparing meals, shopping, doing daily housework, doing laundry, being able to get on a vehicle, being able to use medications, and managing money. 0-8 points are evaluated as "dependent," 9-16 points as "semi-dependent," and 17-24 points as "independent."
Balance and walking assessment | Baseline
  Balance and walking assessment will be assessed with the Tinetti Performance-Oriented Mobility Assessment (POMA). POMA assesses balance ability and walking under 2 main headings. The first 9 questions are about balance, the next 7 questions are about walking. Calculation of the survey score; the total score of the first 9 items gives the balance score, the total score of the next 7 items gives the walking score, and the sum of the balance and walking scores gives the total POMA score. Individuals with a score of 18 and below are considered to have poor balance and walking.
Nutritional assessment | Baseline
  Nutritional assessment will be evaluated with the Mini Nutritional Assessment questionnaire-short form (MNA-SF). MNA-SF consists of 5 subheadings; those with 12-14 points are considered "no risk of malnutrition", those with 8-11 points are considered "at risk of malnutrition" and those with 0-7 points are considered "malnourished".
Frailty | Baseline
  Frailty will be assessed using the Clinical Frailty Scale (CFS). CFS is graded from 1 to 9. The higher the score, the greater the frailty.
Activities of daily living | Baseline
  The assessment of daily living activities will be assessed with the the Barthel Index (BI) scale. BI consists of 10 questions that evaluate feeding, washing, self-care, dressing, defecation control, urinary control, going to the toilet, the ability to get from bed to a wheelchair, mobility status such as walking or being wheelchair dependent, and climbing stairs. 0-20 points are considered as completely dependent, 21-61 points as severely dependent, 62-90 points as moderately dependent, 91-99 points as slightly dependent, and 100 points as completely independent.

CONTACTS AND LOCATIONS:
Overall Officials: Kübra Altunkalem Seydi, MD, Principal Investigator — Sultan 1. Murat State Hospital
Locations (1):
- Sultan 1. Murat State Hospital, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
If requested, the data of the study will be shared by the researchers.